CLINICAL TRIAL: NCT04479098
Title: Effects of Training and Detraining on Body Composition and Inflammatory, Oxidative and Lipid Profiles of Postmenopausal Breast Cancer Survivors Undergoing Tamoxifen Treatment
Brief Title: Effects of Training and Detraining on Postmenopausal Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Igor Moraes Mariano, Principal Investigator, Federal University of Uberlandia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP 57837416.5.0000.5152/2016
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Breast Neoplasm Female
Keywords: Breast Cancer; Immune function; Inflammation; Resistance exercise; Oxidative Stress; Menopause
MeSH Terms: conditions — Breast Neoplasms; Inflammation | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise training (Experimental): Postmenopausal breast cancer survivors undergoing tamoxifen treatment, who will do the evaluations before the beginning and after 12 weeks of exercise training and subsequently 12 weeks of detraining.
  Interventions: Other: Resistance exercise training; Other: Exercise detraining

INTERVENTIONS:
Other: Resistance exercise training — The exercise training program will last 12 weeks, with a frequency of three sessions per week, held on Mondays, Wednesdays, and Fridays. Each session will last approximately 50 minutes. Whenever the maximum number of pre-established repetitions is successfully performed, the intensity will be increased by 5 to 10%. All sessions will be supervised by trained professionals.
Other: Exercise detraining — The exercise detraining will last 12 weeks without exercise.

SUMMARY:
The present study aimed to verify the effects of resistance exercise training and successive detraining on body composition, lipid profile, muscle strength, oxidative stress, and inflammatory markers of postmenopausal breast cancer survivors undergoing tamoxifen treatment.

DETAILED DESCRIPTION:
The present study aimed to verify the effects of 12 weeks of resistance exercise training and successive 12 weeks of detraining on body composition (Body Mass, Body Mass Index, Fat Mass, and Fat-Free Mass), lipid profile (Triglycerides, Total Cholesterol, LDL-Cholesterol, HDL-Cholesterol), muscle strength (1RM test), oxidative stress (Thiobarbituric acid reactive substances,Non-Protein Thiols, Catalase activity, and Superoxide Dismutase), and inflammatory markers (Interferon γ, Tumor Necrosis Factor α, interleukin 6 , Adiponectin, and Interleukin 4) of postmenopausal breast cancer survivors undergoing tamoxifen treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) age between 40 and 65 years; 2) stage 0-IIIA Breast Cancer; 3) submission to axillary lymphadenectomy); 4) completion of chemotherapy and radiation therapy at least 6 months before the study; 5) lack of participation in supervised physical exercise programs in the six months before the beginning of the research; 6) absence of a problem and/or musculoskeletal limitation that would prevent the performance of the proposed exercises; 7) release by a medical professional to participate in the physical training program; 8) residency in Uberlândia

Exclusion Criteria:

* missing more than 20% of the exercise sessions; unable to perform the proposed training protocols; change in drug therapy during the intervention.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in blood biomarkers (pg/mL) | Before and within 72 hours after 12 weeks of exercise training/detraining
  Blood samples will be collected after 8-10 hours overnight fasting directly in evacuated tubes containing separator gel. After centrifugation for 10 min at 3000 rpm, the serum will be separated for immediate analysis or stored at -80 °C for further analysis. Serum levels of IL-4, IL-6, IFN-γ, TNF-α and Adiponectin will be determined by enzyme-linked immunosorbent assays (ELISA) using commercial kits (BD Biosciences, San Jose, CA, USA), according to the manufacturer's instructions, in an Immulite 2000 analyzer (BD Biosciences, San Jose, CA, USA). Expressed in pg/mL.
Changes in blood biomarkers (mmol/L) | Before and within 72 hours after 12 weeks of exercise training/detraining
  Blood samples will be collected after 8-10 hours overnight fasting in evacuated tubes containing separator gel. After 10 min centrifugation at 3000 rpm, the serum will be stored at -80 °C for further analysis. Lipid peroxidation was estimated by determining the serum concentration of thiobarbituric acid reactive substances (TBARS). The TBARS concentration will be obtained by spectrophotometric reading at 535 nm and interpolation in a malondialdehyde calibration curve. Oxidative damage to serum proteins will be estimated by determining the concentration of carbonylated proteins by reading the absorbance at 370 nm and using the molar absorptivity coefficient of 22.000 M-1cm-1. The levels of non-protein thiols will be obtained by the colorimetric method based on the reaction of the sulfhydryl group with 5,5'-dithiobis (2-nitrobenzoic acid) (DTNB). Expressed in mmol/L.
Changes in blood biomarkers (K/gHb.s) | Before and within 72 hours after 12 weeks of exercise training/detraining
  Blood samples will be collected after 8-10 hours overnight fasting directly in evacuated tubes containing separator gel. After centrifugation for 10 min at 3000 rpm, the serum will be separated for immediate analysis or stored at -80 °C for further analysis.Catalase (Cat) activity was evaluated by the ability of this enzyme to convert H2O2 into O2 and H2O. Expressed in K/gHb.s.
Changes in blood biomarkers (U/gHb) | Before and within 72 hours after 12 weeks of exercise training/detraining
  Blood samples will be collected after 8-10 hours overnight fasting directly in evacuated tubes containing separator gel. After centrifugation for 10 min at 3000 rpm, the serum will be separated for immediate analysis or stored at -80 °C for further analysis. The activity of superoxide dismutase (SOD) was evaluated based on their ability to inhibit pyrogallol auto-oxidation and promote a decline in absorbance at 420 nm over time. Expressed in U/gHb.
Changes in blood biomarkers (mg/dL) | Before and within 72 hours after 12 weeks of exercise training/detraining
  Blood samples will be collected after 8-10 hours overnight fasting directly in evacuated tubes containing separator gel. After centrifugation for 10 min at 3000 rpm, the serum will be separated for immediate analysis or stored at -80 °C for further analysis. The serum levels of triglycerides (TGC), total cholesterol (t-C), high-density lipoprotein cholesterol (HDL-C) and low-density lipoprotein cholesterol (LDL-C) will be determined using commercial kits (Labtest, Lagoa Santa, MG, Brazil) in a Technicon RA-XT biochemical analyzer (Bayer, New York, NY, USA). Expressed in mg/dL.

SECONDARY OUTCOMES:
Strength (kg) | Before and within 72 hours after 12 weeks of exercise training/detraining
  The test of one-repetition maximum (1-RM) was adopted to assess muscle strength in all exercises, except for abdominal exercise on the ground, which will be performed only with body mass. Before each test, the subjects will perform a general warm-up (3-5 minutes of light activity), followed by dynamic stretches also for the muscles involved. Then, the participants will perform a specific set of warm-ups that consisted of 8 repetitions with approximately 50% of the estimated load for 1-RM, followed by 3 repetitions with 70% of the estimated load for 1-RM. Subsequently, the loads will be progressively increased until the 1-RM load was found. Rest intervals of approximately 4 to 5 minutes will be inserted between each attempt and the result will be considered valid when performed properly, in a controlled manner, and without assistance from the researchers involved in the assessment. The number of attempts to determine such values will be not more than five. Expressed in kg.
Anthropometry (kg) | Before and within 72 hours after 12 weeks of exercise training/detraining
  Fat mass (FM) and lean mass (LM) will be measured using a tetrapolar bioimpedance analyzer (InBody230™, Seoul, Korea). Expressed in kg.
Anthropometry (%) | Before and within 72 hours after 12 weeks of exercise training/detraining
  Fat mass percentage (BF%) will be measured using a tetrapolar bioimpedance analyzer (InBody230™, Seoul, Korea).
Anthropometry (kg/m²) | Before and within 72 hours after 12 weeks of exercise training/detraining
  Height was measured in a stadiometer with 0.1 cm accuracy and total body mass was measured using a balance with 0.1 kg accuracy. Body mass index will be calculated using the formula: body mass/height². Expressed in kg/m².

CONTACTS AND LOCATIONS:
Locations (1):
- Guilherme Morais Puga, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided